CLINICAL TRIAL: NCT02270931
Title: A Prospective Longitudinal Study of CA 15-3 as an Aid in Monitoring Recurrence or Progressive Disease in Patients With Breast Cancer
Brief Title: A Prospective Longitudinal Breast Cancer Study
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-69
Record Dates: First submitted 2014-10-02; First posted 2014-10-22 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CA 15-3 Assay — Physicians use the CA 15-3 test result to manage their patients

SUMMARY:
The purpose of this study is to obtain sufficient specimens and correlating clinical data from a well-controlled prospective clinical trial collecting longitudinal specimens from subjects diagnosed with any stage of breast cancer.

DETAILED DESCRIPTION:
The study objectives are described below:

1. Obtain serum and plasma specimens longitudinally collected from a minimum of 130 subjects diagnosed with breast cancer and are about to or are currently undergoing treatment and follow-up. Specimens will be used to evaluate CA 15-3 assays, currently under development, as an aid for monitoring recurrence or progressive disease.
2. To store any remaining specimens for use in future cancer research and to evaluate as yet undetermined biomarkers for the development of IVDs, including additional CA 15-3 assays, for monitoring the course of disease and therapy in subjects diagnosed with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age≥ 18 years
* Histologic/pathologic confirmation of breast cancer
* Any stage of disease: Newly diagnosed, stable, disease progression, surveillance
* Any treatment time point: Treatment naïve, currently receiving or completed therapy for breast cancer including active monitoring.
* Individuals with a history of malignant disease other than breast cancer that was resected greater than 5 years ago and are currently in remission are eligible.
* Able to understand and willing to provide informed consent

Exclusion Criteria:

* Males and females, age <18 years
* No histologic/pathologic confirmation of breast cancer
* Any concurrent malignancy other than basal or squamous cell skin cancers, in-situ cervical cancer, or breast cancer.
* Treatment plan with fewer than three visits expected in 3 years' time
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 130 subjects will be enrolled in this study. Women and men greater than or equal to 18 years of age with a histologically/pathologically confirmed diagnosis of breast cancer and a minimum of three serial blood draws collected at disease evaluation time points, as determined by the treating physician's standard of care, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2014-05; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Measure CA 15-3 in Breast Cancer Patients | 3 years
  130 patients with Recurrence or Progressive Breast Cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, Study Director — Fujirebio Diagnostics, Inc.
Locations (3):
- United States (3):
  - Jane Skelton, MD, Boca Raton, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - New Hanover Regional Medical Center, Wilmington, North Carolina